CLINICAL TRIAL: NCT03119168
Title: The Effect Of Adding High Dose Simethicone To A Standard Polyethylene Glycol Preparation On Adenoma Detection Rate During Screening Colonoscopy: A Randomized Controlled Pilot Trial
Brief Title: Effect of Simethicone on Screening Colonoscopy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Texas Tech University Health Sciences Center, El Paso (Other)
Responsible Party: Principal Investigator, Antonio Mendoza-Ladd, Assistant Professor of Medicine, Texas Tech University Health Sciences Center, El Paso
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: E17034
Record Dates: First submitted 2017-04-10; First posted 2017-04-18 (Actual); Results first posted 2019-06-05 (Actual); Last update posted 2019-06-05 (Actual); Status verified 2019-06

CONDITIONS: Adenoma Colon
Keywords: screening; adenoma detection rate; simethicone
MeSH Terms: interventions — Simethicone; alginate-polyethylene glycol acrylate

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Simethicone solution + Polyethylenglycol (Experimental): This arm of the study will include the patients assigned to take simethicone solution with their colon preparations ( 4L Polyethyleneglycol)
  Interventions: Drug: Simethicone Solution
- Polyethylenglycol (Active Comparator): This arm of the study will include the patients assigned to take a regular bowel preparation (4L Polyethylenglycol)
  Interventions: Other: Polyethylenglycol

INTERVENTIONS:
Drug: Simethicone Solution — Patients will be assigned randomly to take Simethicone Solution plus polyethylenglycol
  Other Names: mylicon
  Arms: Simethicone solution + Polyethylenglycol
Other: Polyethylenglycol — Patients in this arm will be randomly assigned to take polyethylenglycol as their regular bowel preparation
  Arms: Polyethylenglycol

SUMMARY:
This study is evaluating the effect of adding a high dose of simethicone to the standard polyethylene glycol preparation for screening colonoscopy in the quality of the preparation , adenoma detection rate and withdrawal times.

DETAILED DESCRIPTION:
A proper bowel preparation is key to a thorough and safe colonoscopy. Several factors affect the mucosal visualization during colonoscopy, and consequently the quality of such evaluation. Undoubtedly, this can have unfavorable implications like missed lesions. One of the most commonly encountered scenarios is the presence of multiple bubbles that interfere with mucosal visualization. When this occurs, simethicone (an antifoam agent used to reduce bloating when ingested orally) is injected through the colonoscope to eliminate the bubbles and get a clear view of the mucosa. A few studies have used oral simethicone in conjunction with oral preparation agents (PEG, magnesium citrate, sodium phosphate) in an attempt to improve the quality of the preparation. Unfortunately these studies have not used the exact same preparation agent with and without simethicone, making it difficult to draw conclusions on its efficacy. However, it is important to understand that simethicone is not intended to decrease the amount of stool in the colon, and it's purpose is to decrease the amount of bubbles interfering with the visualization of the mucosa provided that there is no stool present . Furthermore, it is unclear if adding simethicone to a standard bowel preparation makes a significant difference in key aspects of screening colonoscopy such as adenoma detection rate or withdrawal times. This prospective randomized controlled, observer blinded study at Texas Tech University Health Sciences Center in El Paso, aims at studying the effect of simethicone on the overall colon preparation as well as on adenoma detection rate and withdrawal times.

ELIGIBILITY:
Inclusion Criteria:

1. Patients between the ages of 30-80 scheduled for screening colonoscopy.
2. Male and female patients
3. Ambulatory patients
4. Signed informed consent form

Exclusion Criteria:

1. Previous colonic surgery
2. Patient with mental/physical condition that impairs oral ingestion of preparation
3. Allergy or hypersensitivity to simethicone
4. Patients with limited mobility (bedridden patients)
5. Patients with gastrointestinal obstruction
6. Patients with gastroparesis

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 268 (Actual)
Dates: Start 2017-03-15 (Actual); Primary Completion 2019-04-10 (Actual); Study Completion 2019-04-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Antonio H Mendoza-Ladd, MD, Principal Investigator — Texas Tech University Health Sciences Center, El Paso
Locations (1):
- Texas Tech university Health Sciences Center El Paso, El Paso, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Park JJ, Lee SK, Jang JY, Kim HJ, Kim NH. The effectiveness of simethicone in improving visibility during colonoscopy. Hepatogastroenterology. 2009 Sep-Oct;56(94-95):1321-5. PMID 19950784
- [Background] Yoo IK, Jeen YT, Kang SH, Lee JH, Kim SH, Lee JM, Choi HS, Kim ES, Keum B, Chun HJ, Lee HS, Kim CD. Improving of bowel cleansing effect for polyethylene glycol with ascorbic acid using simethicone: A randomized controlled trial. Medicine (Baltimore). 2016 Jul;95(28):e4163. doi: 10.1097/MD.0000000000004163. PMID 27428209
- [Result] Rex DK, Petrini JL, Baron TH, Chak A, Cohen J, Deal SE, Hoffman B, Jacobson BC, Mergener K, Petersen BT, Safdi MA, Faigel DO, Pike IM. Quality indicators for colonoscopy. Gastrointest Endosc. 2006 Apr;63(4 Suppl):S16-28. doi: 10.1016/j.gie.2006.02.021. No abstract available. PMID 16564908
- [Result] Hassan C, Fuccio L, Bruno M, Pagano N, Spada C, Carrara S, Giordanino C, Rondonotti E, Curcio G, Dulbecco P, Fabbri C, Della Casa D, Maiero S, Simone A, Iacopini F, Feliciangeli G, Manes G, Rinaldi A, Zullo A, Rogai F, Repici A. A predictive model identifies patients most likely to have inadequate bowel preparation for colonoscopy. Clin Gastroenterol Hepatol. 2012 May;10(5):501-6. doi: 10.1016/j.cgh.2011.12.037. Epub 2012 Jan 10. PMID 22239959
- [Derived] Moraveji S, Casner N, Bashashati M, Garcia C, Dwivedi A, Zuckerman MJ, Carrion A, Ladd AM. The role of oral simethicone on the adenoma detection rate and other quality indicators of screening colonoscopy: a randomized, controlled, observer-blinded clinical trial. Gastrointest Endosc. 2019 Jul;90(1):141-149. doi: 10.1016/j.gie.2019.03.018. Epub 2019 Mar 26. PMID 30926430

RESULTS

PARTICIPANT FLOW:
Groups:
- Simethicone Solution + Polyethylenglycol: This arm of the study will include the patients assigned to take simethicone solution with their colon preparation (4L Polyethylenglycol)
  Simethicone Solution: Patients will be assigned randomly to take Simethicone Solution plus 4 L of polyethylenglycol
- Polyethylenglycol: This arm of the study will include the patients assigned to take a regular bowel preparation with 4L Polyethylenglycol
  Polyethylenglycol: All patients were assigned to take 4L polyethylenglycol as their regular bowel preparation
Period: Overall Study
Arm/Group | Simethicone Solution + Polyethylenglycol | Polyethylenglycol
Started | 129 | 139
Completed | 129 | 139
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Simethicone Solution + Polyethylenglycol: This arm of the study will include the patients assigned to take simethicone solution with their colon preparations
  Simethicone Solution: Patients will be assigned randomly to take Simethicone Solution plus polyethylenglycol
- Polyethylenglycol: This arm of the study will include the patients assigned to take a regular bowel preparation with Polyethylenglycol
  Polyethylenglycol: Patients in this arm will be randomly assigned to take polyethylenglycol as their regular bowel preparation
- Total: Total of all reporting groups
Arm/Group | Simethicone Solution + Polyethylenglycol | Polyethylenglycol | Total
Number analyzed (Participants) | 129 | 139 | 268
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.3 (7.55) | 57 (6.02) | 57 (6.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 81 | 92 | 173
  Male | 48 | 47 | 95
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic | 111 | 124 | 235
  Non Hispanic | 18 | 15 | 33
Region of Enrollment [Number; unit: participants]
  United States | 129 | 139 | 268
Count of participants [Count of Participants; unit: Participants] | 129 | 139 | 268

OUTCOME MEASURES:

1. Primary Outcome: Adenoma Detection Rate
Description: The number of adenomatous polyps removed at colonoscopy
Time Frame: 25 minutes
Measure: Number; unit: adenomas
Arm/Group | Simethicone Solution + Polyethylenglycol | Polyethylenglycol
Number analyzed (Participants) | 129 | 139
adenomas | 43 | 54

2. Secondary Outcome: Withdrawal Times
Description: Amount spent withdrawing the scope during the colonoscopy
Time Frame: 6-10 minutes
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Simethicone Solution + Polyethylenglycol | Polyethylenglycol
Number analyzed (Participants) | 129 | 139
seconds | 395.7 (69.2) | 399 (76.7)

3. Secondary Outcome: Colon Preparation
Description: Boston Bowel Preparation Scale (BBPS): scale that rates the quality of the colon preparation based on the amount of stool present. 0:solid stool that cannot be cleared; 1:areas not well seen due to residual stool and/or opaque liquid; 2:small fragments of stool and/or opaque liquid, but mucosa seen well; 3:no residual stool or opaque liquid seen. Score determined by adding the score of each individual segment of the colon (right side, transverse and left side). Scores range from 0 to 3 in each segment, therefore, a total composite score ranges from 0 (poor) to 9 (excellent).
  Bubble Score (BS): scale that rates the amount of bubbles present in the colon. 0:no or minimal bubbles; 1:bubbles covering up to half the luminal diameter; 2:bubbles covering the circumference of the lumen; 3:bubbles filling the entire lumen. Score determined the same way as BBPS score but in this case a total score of 0 is excellent and 9 is poor.
Time Frame: 25 minutes
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Simethicone Solution + Polyethylenglycol | Polyethylenglycol
Number analyzed (Participants) | 129 | 139
score on a scale
  Boston Bowel Preparation Scale | 8.9 (0.4) | 8.9 (0.4)
  Bubble Scale | 0.1 (0.2) | 2.1 (2.1)

4. Secondary Outcome: Intraprocedural Use of Simethicone
Description: The number of colonoscopies during which the endoscopist requested simethicone to be flushed through the endoscope.
Time Frame: 6-10 minutes
Measure: Number; unit: colonoscopies
Groups:
- Simethicone Solution + Polyethylenglycol; Polyethylenglycol: The number of colonoscopies during which the endoscopist requested simethicone to be flushed through the endoscope
Arm/Group | Simethicone Solution + Polyethylenglycol | Polyethylenglycol
Number analyzed (Participants) | 129 | 139
colonoscopies | 2 | 68

ADVERSE EVENTS:
Time Frame: 60 minutes
Groups:
- Simethicone Solution + Polyethylenglycol: Simethicone solution + Polyethylenglycol were received as a bowel prep regimen
- Polyethylenglycol: Polyethylenglycol was received as a bowel prep regimen
Arm/Group | Simethicone Solution + Polyethylenglycol | Polyethylenglycol
All-Cause Mortality (participants affected / at risk) | 0/129 | 0/139
Serious Adverse Events (participants affected / at risk) | 0/129 | 0/139
Other Adverse Events (participants affected / at risk) | 0/129 | 0/139

LIMITATIONS AND CAVEATS:
The study was done at our hospital setting, generalizability can be examined in larger studies

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-01-10): https://cdn.clinicaltrials.gov/large-docs/68/NCT03119168/Prot_SAP_000.pdf
  • Informed Consent Form (2018-08-02): https://cdn.clinicaltrials.gov/large-docs/68/NCT03119168/ICF_001.pdf